CLINICAL TRIAL: NCT01014689
Title: Efficacy and Safety Comparison of Epiduo Gel Associated With Lymecycline 300 mg Capsules Versus Epiduo Vehicle Gel Associated With Lymecycline 300 mg Capsules in the Treatment of Moderate to Severe Acne Vulgaris
Brief Title: Comparison of Epiduo Associated With Lymecycline Versus Epiduo Vehicle Associated With Lymecycline in Acne Vulgaris
Acronym: TEAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.03.SPR.29080
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2012-04

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Lymecycline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adapalene 0.1% / BPO 2.5% gel (Active Comparator)
  Interventions: Drug: Adapalene/ BPO gel with Lymecycline capsules
- Adapalene 0.1% / BPO 2.5% Vehicle Gel (Placebo Comparator)
  Interventions: Drug: Adapalene/ BPO vehicle gel with Lymecycline capsules

INTERVENTIONS:
Drug: Adapalene/ BPO gel with Lymecycline capsules — Gel: Topical to the face, once daily in the evening Capsule: 1 capsule once daily in the morning
  Other Names: Adapalene/BPO with Lymecycline
  Arms: Adapalene 0.1% / BPO 2.5% gel
Drug: Adapalene/ BPO vehicle gel with Lymecycline capsules — Gel: Topical to the face, once daily in the evening Capsule: 1 capsule once daily in the morning
  Other Names: Adapalene/BPO vehicle with Lymecycline
  Arms: Adapalene 0.1% / BPO 2.5% Vehicle Gel

SUMMARY:
Randomized, controlled, multi-center, double-blind, parallel-group comparison study in Subjects with moderate to severe acne vulgaris on the face.

The purpose of this study is to demonstrate the efficacy of Adapalene 0.1% / Benzoyl Peroxide (BPO) 2.5% Gel associated with Lymecycline 300mg Capsules compared to Adapalene 0.1% /Benzoyl Peroxide 2.5% Vehicle Gel associated with Lymecycline 300mg Capsules, in the treatment of moderate to severe acne vulgaris.

The safety of the two treatment regimens will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Subjects of any race, aged 12 to 35 years inclusive,
2. Subjects with moderate to severe facial acne vulgaris (Investigator's Global Assessment score of 3 or 4),

Exclusion Criteria:

1. Subjects with more than 3 nodules or cysts on the face
2. Subjects with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.),
3. Subjects with a wash-out period for topical treatment on the face less than: Corticosteroids, antibiotics, antibacterials, antiseptics, retinoids, other anti-inflammatory drugs or other acne treatments (2 weeks), Zinc containing drugs (1 week), Phototherapy devices for acne and cosmetic procedures (1 week)
4. Subjects with a wash-out period for systemic treatment less than:Acne therapy containing zinc (4 weeks), Corticosteroids, antibiotics (4 weeks), Other acne treatments (6 months), Ciproterone acetate / Chlormadinone acetate (6 months), Spironolactone / Drospirenone (3 months)
5. Subjects with impaired hepatic (ALT/AST > 3xULN and bilirubin > 1.5xULN) or renal (creatinine clearance greater than 60 ml/min) functions based on a blood sample,
6. Subjects with known intolerance to lactose,

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 378 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Paliargues, Study Director — Galderma R&D
Locations (28):
- Australia (4):
  - Galderma Investigator site, Canberra
  - Galderma Investigator site, Kogarah
  - Galderma Investigator site, Melbourne
  - Galderma Investigator site, Sydney
- Belgium (3):
  - Galderma Investigator site, Brussels
  - Galderma Investigator site, Ghent
  - Galderma Investigator site, Leuven
- Brazil (2):
  - Galderma Investigator site, Belo Horizonte
  - Galderma Investigator site, São Paulo
- France (6):
  - Galderma Investigator site, Bordeaux
  - Galderma Investigator site, Cannes
  - Galderma Investigator site, Martigues
  - Galderma Investigator site, Nantes
  - Galderma Investigator site, Pantin
  - Galderma Investigator site, Pierre-Bénite
- Germany (3):
  - Galderma Investigator site, Cuxhaven
  - Galderma Investigator site, Darmstadt
  - Galderma Investigator site, Frankfurt
- Italy (2):
  - Galderma Investigator site, Catania
  - Galderma Investigator site, Ferrara
- Mexico (4):
  - Galderma Investigator site, Mexico City
  - Galderma Investigator site, Monterrey
  - Galderma Investigator site, Tlalnepantla
  - Galderma Investigator site, Zapopan
- Galderma Investigator site, Lodz, Poland
- Sweden (3):
  - Galderma Investigator site, Eskilstuna
  - Galderma Investigator site, Farsta
  - Galderma Investigator site, Hägersten

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 14/08/2009 to 21/01/2010 Type of location: hospital, private hospital and private practice.
Groups:
- Adapalene 0.1% / BPO 2.5% Gel + Lymecycline; Adapalene 0.1% / BPO 2.5% Vehicle Gel + Lymecycline: Gel applied once daily in the evening during 12 weeks Lymecycline 300mg taken once daily in the morning during 12 weeks
Period: Overall Study
Arm/Group | Adapalene 0.1% / BPO 2.5% Gel + Lymecycline | Adapalene 0.1% / BPO 2.5% Vehicle Gel + Lymecycline
Started | 191 | 187
Completed | 178 | 174
Not Completed | 13 | 13
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 3 | 7
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapalene 0.1% / BPO 2.5% Gel + Lymecycline | Adapalene 0.1% / BPO 2.5% Vehicle Gel + Lymecycline | Total
Number analyzed (Participants) | 191 | 187 | 378
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 113 | 102 | 215
  Between 18 and 65 years | 78 | 85 | 163
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.6 (4.7) | 19.1 (4.6) | 18.9 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 78 | 169
  Male | 100 | 109 | 209
Region of Enrollment [Number; unit: participants]
  France | 26 | 25 | 51
  Mexico | 52 | 52 | 104
  Brazil | 18 | 17 | 35
  Poland | 16 | 16 | 32
  Belgium | 14 | 13 | 27
  Australia | 15 | 18 | 33
  Germany | 18 | 17 | 35
  Italy | 14 | 14 | 28
  Sweden | 18 | 15 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Lesion Count
Description: Percent change from Baseline in Total Lesion count (sum of Non-Inflammatory and Inflammatory lesions) at Week 12.
Time Frame: Baseline and Week 12
Population: Intention to treat - Last observation carried forward
Measure: Median (Full Range); unit: percent of change
Arm/Group | Adapalene 0.1% / BPO 2.5% Gel + Lymecycline | Adapalene 0.1% / BPO 2.5% Vehicle Gel + Lymecycline
Number analyzed (Participants) | 191 | 187
percent of change | -74.1 [-100 to 7.7] | -56.8 [-97.8 to 73.2]

2. Secondary Outcome: Success Rate on the Investigator's Global Assessment (IGA) at Week 12
Description: Percentage of Subjects "Clear" or "Almost Clear" on 6-point IGA scale(0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe and 5=very severe) at Week 12.
Time Frame: Baseline and Week 12
Population: Intention To treat - Last Observation Carried Forward
Measure: Number; unit: percent of subjects
Arm/Group | Adapalene 0.1% / BPO 2.5% Gel + Lymecycline | Adapalene 0.1% / BPO 2.5% Vehicle Gel + Lymecycline
Number analyzed (Participants) | 191 | 187
percent of subjects | 47.6 | 33.7

ADVERSE EVENTS:
Time Frame: 12 weeks.
Description: All clinical medical events, occured after Subject's consent signed and during the study, whether observed by the Investigator or reported by the Subject and whether or not thought to be product- or study procedure-related were considered adverse events and collected.
Arm/Group | Adapalene 0.1% / BPO 2.5% Gel + Lymecycline | Adapalene 0.1% / BPO 2.5% Vehicle Gel + Lymecycline
Serious Adverse Events (participants affected / at risk) | 0/191 | 0/187
Other Adverse Events (participants affected / at risk) | 25/191 | 26/187
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene 0.1% / BPO 2.5% Gel + Lymecycline (N=191) | Adapalene 0.1% / BPO 2.5% Vehicle Gel + Lymecycline (N=187)
HEADACHE (Nervous system disorders) | 12 (19) | 17 (23)
NASOPHARYNGITIS (Infections and infestations) | 14 (15) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreement in full force and effect for a period of 10 years.